CLINICAL TRIAL: NCT06504433
Title: The Natural History of Mitochondrial Diseases
Status: Recruiting | Type: Observational
Sponsor: Neuroscience Research Australia (Other)
Responsible Party: Sponsor
Other Study IDs: 2024_ETH00044
Record Dates: First submitted 2024-07-11; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Mitochondrial Diseases; Neurological Diseases or Conditions; Parkinson Disease; Genetic Disease
MeSH Terms: conditions — Mitochondrial Diseases; Parkinson Disease; Genetic Diseases, Inborn | interventions — Sequence Deletion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — MITO and control Participants (asymptomatic, unaffected family members, or patients with non-MITO movement disorder), the following biospecimens will be collected to form the biobank for DNA extraction, biomarker and heteroplasmy analysis:
  1. Whole blood collection (60ml every 6 months ii. Plasma and serum iii. PBMCs will be extracted for transcriptomics, proteomics and possible cell line iv. development
  2. Skin biopsies will be used to create fibroblast cells
  3. Hair follicles
  4. Urine and urinary epithelial cells every 6 months will be used for autofluorescence analysis, metabolomics, biomarker development and DNA extraction
  5. Saliva/Buccal cells
  6. Stool will be collected, via a home collection kit, every 6 to 12 months, for microbiome analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MITO participants/patients: 400 MITO patients will be observed over 10 years and having a confirmed variant/deletion in either nuclear or mitochondrial genes involved in the mitochondrial respiratory chain, or patients meeting the clinical diagnostic criteria for MITO using consensus scoring systems such as the Walker Criteria, or the Nijmegen criteria
  Interventions: Diagnostic Test: Confirmed variant/deletion in either nuclear or mitochondrial genes involved in the mitochondrial respiratory chain
- Patients with a clinically confirmed non-MITO neuromuscular disorder: The study will form a 10-year, longitudinal, non-randomised, retrospective, and prospective, observational study of patients with MITO using controls who may be:
  * asymptomatic biological relatives of MITO participants/patients
  * patients with a clinically confirmed non-MITO neuromuscular disorder, or
  Interventions: Diagnostic Test: Confirmed variant/deletion in either nuclear or mitochondrial genes involved in the mitochondrial respiratory chain
- Age and gender-matched healthy controls.: Age/gender-matched healthy controls will be recruited from the NeuRA database of volunteers
  Interventions: Diagnostic Test: Confirmed variant/deletion in either nuclear or mitochondrial genes involved in the mitochondrial respiratory chain

INTERVENTIONS:
Diagnostic Test: Confirmed variant/deletion in either nuclear or mitochondrial genes involved in the mitochondrial respiratory chain — This is a 10-year, longitudinal, non-randomised, retrospective and prospective, observational study that will be used to characterise the natural history of primary mitochondrial disease (MITO) in 400 participants and their asymptomatic family members (with no genetic risk), non-MITO healthy controls (100 participants) and form a biobank that can be used in future research using separate ethics approved protocols to identify biomarkers of disease onset and progression.

SUMMARY:
The Natural History of Mitochondrial (MITO) Diseases (a longitudinal study observing the natural history of mitochondrial diseases)

The goal of this observational study (non-randomised retrospective and prospective) is to fully characterise primary MITO disease; that includes both sexes/genders, over 18 years of age and healthy volunteers]. The main question[s] it aims to answer is to:

• better characterise MITO phenotypes (organ involvement, severity, progression) and collect biospecimens to create a biobank that can be used for future biomarker discovery to improve early diagnosis, prognostication and management of mitochondrial disease.

The study will be a longitudinal, retrospective, prospective, observational study of participants (400) with confirmed MITO and relevant controls followed for up to 10 years. Data will be collected at regularly scheduled standard-of-care (SOC), 6 to 12 monthly appointments.

The 100 control participants will therefore be comprised of (i) unaffected asymptomatic family members of MITO participants with no genetic risk; (ii) participants with non-MITO movement disorders that are not classified as MITO by their clinical presentation and genetic tests (for example Parkinson's disease) and/or (iii) age-matched healthy controls recruited from the NeuRA database of volunteers.

Demographic data, medical history, biochemical, histological, genetic, social and other clinical SOC data will be collected. Additionally, seizure and migraine frequency in participants who experience these, will be collected and a quality-of-life questionnaire (SF-12v2), as part of the validated neurological assessment using the Newcastle Mitochondrial Disease Adult Scale (NMDAS).

DETAILED DESCRIPTION:
Primary Mitochondrial Disease (MITO) is a serious and debilitating condition, often multi-systemic and requiring life-long monitoring and treatment of symptoms to reduce the risk of life-threatening episodes, metabolic crises, or acute illness. Although rare, MITO is the most common group of inherited metabolic diseases and is associated with abnormalities of the mitochondrial respiratory chain, which carries out oxidative phosphorylation to produce ATP (Gorman et al. 2016).

In adults, MITO is often a progressive multisystem disorder, with frequent, long-term monitoring and symptom management required to reduce the risk of an acute illness, and/or other life-threatening episodes and metabolic crises

Given that mtDNA mutations are typically transmitted through the maternal line, paternally related family members are not at risk and will represent asymptomatic controls. In sporadic cases such as chronic progressive external ophthalmoplegia (CPEO) that are typically caused by sporadic mtDNA deletions, family members are not at risk of carrying the disorder, and thus can act as family member controls. Similarly, those family members of participants with a nuclear DNA mutation such as autosomal dominant mitochondrial disease (e.g., OPA1 gene), and who do not carry the affected gene are also suitable asymptomatic controls.

This study will establish the AMDC Clinical Registry at NeuRA. Patients with confirmed MITO (the presence of pathogenic nuclear or mitochondrial DNA variants/deletion) and control participants that can include: biological relatives of MITO participants with no clinical disease and no genetic risk; participants with a clinically confirmed non-MITO neurologic disorder or age and gender-matched healthy controls followed over at least 120 months (10) years.

Study data will include detailed medical and social history, summary of clinical presentation and clinical social history collected through diaries or on clinical review; neurological examination findings; results of investigations performed as standard of care, including laboratory findings through blood tests, imaging studies, cardiac investigations, gastrointestinal transit studies, neurophysiological studies, and analysis of archived muscle and/or skin biopsies.

Individuals of any age with confirmed MITO that requires the presence of pathogenic nuclear or mitochondrial DNA variants/deletion. Control participants (100) may fall into one of three categories: asymptomatic relatives of confirmed MITO patients (those with no genetic risk); patients with clinically confirmed non-MITO neurological disorders; or age and gender-matched healthy controls.

If genetic mutations are not demonstrated, MITO can be diagnosed using clinical diagnostic criteria, including the Walker Criteria, or the Nijmegen criteria (consensus mitochondrial disease criteria scoring system).

All patients must agree to participate in the Australian Mitochondrial Disease Centre (AMDC) Clinical Registry and donate, at a minimum a blood sample, for the prospective biobank for the collection and storage of biological samples for future use.

Overall, individual disease courses in MITO range from slow to more rapid progressive decline, to stepwise deterioration often attributable to metabolic events, eventuating as a potentially fatal disease. To further complicate these already immense diagnostic and prognostic challenges, external or environmental factors such as toxins, inflammation, nutrition, the microbiome, and the natural aging process, are now being postulated to additionally influence the onset, organ involvement, severity, and progression of disease, although this is poorly understood.

MITO is a vastly heterogeneous disease, and a genetic diagnosis does not necessarily nor comprehensively inform the clinician how the disease will manifest clinically in an individual. A deeper understanding of MITO's natural history and its associated biomarkers will instead provide the clinician with the necessary tools and a greater understanding that optimises patient care. Additionally, it will allow for more accurate:

* screening of patients and when to apply mitochondrial genomic testing,
* prediction of disease severity and prognosis,
* matching of clinical presentations to genotypes,
* monitoring for symptomatic and metabolic changes to minimise/prevent potential crises,
* utilisation of appropriate management plans their effectiveness assessment,
* application of available targeted treatments (and clinical trials), and
* application of preventative strategies such as mitochondrial donation techniques.

By collecting the clinically relevant data of each genetically diagnosed patient, the study will map and identify factors that influence disease, to assist not only current NeuRA clinicians but future clinicians in the management of MITO patients. Biospecimens will be collected to form the Australian Mitochondrial Disease Centre (AMCD) biobank that will facilitate separate and future biomarker discovery research, important for the assessment of organ involvement, disease severity, and responses to therapies. With the benefits of earlier diagnoses, improved patient care and health outcomes, and aiding drug/treatment discovery.

In this longitudinal study, we aim to further define existing and identify the different MITO phenotypes; examine possible associations between specific events in the medical history of the patient; identify correlations between the signs and symptoms of MITO presentations and disease severity, prognostic indicators, and survival; and create an informative biobank. One that can be accessed for future use in ethically approved protocols, and where biospecimens can be reassessed to identify precise mitochondrial biomarkers that aid a timelier MITO diagnosis or prediction of disease progression. Clinical symptoms will also be correlated with environmental factors such as medications, and physical exercise to provide an improved understanding of how treatments, lifestyle, and dietary interventions impact the clinical course of MITO.

Overall Aim: To perform a longitudinal study of MITO over 10 years and create a clinical database to examine possible associations between clinical features, disease phenotypes and disease progression in MITO participants and relevant controls. Various biospecimens will be collected to form a 'biobank' that will facilitate MITO biomarker research and that can be accessed using ethics-approved protocols for future research

Project outcomes This study will establish the AMDC Clinical 'Biobank' repository. Patients with MITO and their asymptomatic relatives (with no genetic risk) will be followed for at least 10 years with biospecimen collection to form a Biobank that will facilitate MITO biomarker research. The data generated may identify triggers of clinical symptoms and associations between clinical and environmental parameters. Future research studies using ethics-approved protocols to access biospecimens in the biobank will facilitate MITO biomarker research that would allow earlier diagnosis of MITO, identify organ involvement, track disease progression to help with prognostication and improve disease management.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical and/or genetically confirmed diagnosis of MITO.
2. Individuals > 18 years of age, managed by a specialist neurologist, with confirmed MITO
3. Control participants will comprise asymptomatic relatives of confirmed MITO patients with no clinical or genetic evidence of MITO; clinically confirmed non-MITO movement disease controls (from other clinics at NeuRA) or age/gender-matched healthy participants.

Exclusion Criteria:

* • Those participants who do NOT match the inclusion criteria above

  * Not willing to participate in the AMDC Clinical Registry
  * Not willing to undergo genetic testing
  * Not willing to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants (at least 400) with confirmed MITO (on genetic/clinical grounds) will be recruited into this study through NeuRA, Randwick, NSW by CI/CPI Professor Carolyn Sue AM FAHMS.
  The study will recruit 100 control participants who may be:
  i. age and gender-matched healthy controls from the NeuRA database of volunteers; ii. asymptomatic relatives of MITO participants or iii. non-MITO movement disorder controls recruited from other clinics at NeuRA.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2029-05-07 (Estimated); Study Completion 2034-05-07 (Estimated)

PRIMARY OUTCOMES:
Descriptive measures: The natural history of mitochondrial disease | 10 years
  The primary outcome measure is the creation of a clinical database and biospecimen repository (biobank) with medical, health and lifestyle data to characterise the natural history of mitochondrial disease for each MITO patient. Data will be stratified by disease genotype, phenotype, age of onset, sequence and timing of major symptom onset, severity and progression of organ involvement and symptom progression, to identify any associations between parameters.

SECONDARY OUTCOMES:
The natural history of mitochondrial disease | 10 years
  The secondary outcomes will be the creation of a biospecimen repository (biobank) for biomarker discovery research to improve diagnosis, and disease progression and identify possible treatments. External collaborators, using ethics-approved protocols, may apply to access the biobank to analyse biospecimens for biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn M Sue, MBBS, Principal Investigator — Kinghorn Chair, Neuroscience Research Australia
Locations (1):
- Neuroscience Research Australia, Randwick, New South Wales, Australia

REFERENCES:
- [Background] Davis RL, Liang C, Sue CM. A comparison of current serum biomarkers as diagnostic indicators of mitochondrial diseases. Neurology. 2016 May 24;86(21):2010-5. doi: 10.1212/WNL.0000000000002705. Epub 2016 Apr 27. PMID 27164684
- [Background] Davis RL, Liang C, Sue CM. Mitochondrial diseases. Handb Clin Neurol. 2018;147:125-141. doi: 10.1016/B978-0-444-63233-3.00010-5. PMID 29325608
- [Background] Sue CM, Balasubramaniam S, Bratkovic D, Bonifant C, Christodoulou J, Coman D, Crawley K, Edema-Hildebrand F, Ellaway C, Ghaoui R, Kava M, Kearns LS, Lee J, Liang C, Mackey DA, Murray S, Needham M, Rius R, Russell J, Smith NJC, Thyagarajan D, Wools C. Patient care standards for primary mitochondrial disease in Australia: an Australian adaptation of the Mitochondrial Medicine Society recommendations. Intern Med J. 2022 Jan;52(1):110-120. doi: 10.1111/imj.15505. Epub 2021 Nov 19. PMID 34505344